CLINICAL TRIAL: NCT06697678
Title: Development and Validation of a Risk Prediction Model for Severe Autoimmune Encephalitis
Brief Title: Risk Prediction Model for Severe Autoimmune Encephalitis
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: AE
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Severe Autoimmune Encephalitis
Keywords: severe autoimmune encephalitis; prediction model; plasma exchange therapy; plasma adsorption therapy; targeted immunotherapy
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with severe autoimmune encephalitis: No intervention
  Interventions: Other: No Intervention: Observational Cohort
- patients with non-severe autoimmune encephalitis
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
A prospective study aims to establish a multicenter clinical diagnosis and treatment database for patients with autoimmune encephalitis (AE). The study will analyze the characteristics of disease progression, changes in immune-inflammatory markers, immunotherapy regimens, and patient outcomes. It seeks to identify clinical indicators for the early recognition of severe AE patients, develop and validate a predictive model for severe AE, and explore effective treatment strategies to rapidly control disease progression during the acute phase of severe AE.

DETAILED DESCRIPTION:
To develop and validate a predictive model for severe autoimmune encephalitis (AE), a prospective multicenter study will be conducted. Clinical data of hospitalized AE patients will be collected consecutively, and a multicenter integrated database will be established. This database will include information on the characteristics of disease progression, changes in blood and cerebrospinal fluid immune-inflammatory markers, specific immunotherapy regimens, patient outcomes, and long-term prognoses. The study will analyze the clinical and immunological characteristics of AE patients, identify clinical indicators for early recognition of severe AE, and develop and validate a predictive model for severe AE. Additionally, the study will evaluate the efficacy of early plasma exchange/plasma adsorption therapy and targeted immunotherapy on AE outcomes and long-term prognosis, aiming to explore effective treatment strategies for rapidly controlling disease progression in the acute phase of severe AE.

ELIGIBILITY:
Inclusion Criteria:

* age 14-80 years
* no restriction on gender
* meets the diagnostic criteria for confirmed AE, with a clearly identified pathogenic antibody
* within 3 months of AE
* patients voluntarily sign the informed consent form; if unable to express their will or sign, the consent form can be signed by a close relative on their behalf

Exclusion Criteria:

* no lumbar puncture performed for CSF antibody testing
* did not receive immunotherapy
* pre-onset modified Rankin Scale (mRS) score ≥3

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnostic criteria for autoimmune encephalitis (AE) patients (all four criteria must be met): A. clinical Presentation: acute or subacute onset (<3 months) with one or more neurological or psychiatric symptoms or clinical syndromes: a. limbic system symptoms b. encephalitis syndrome c. basal ganglia and/or diencephalon/hypothalamus involvement d. psychiatric disorders. B. auxiliary tests: presence of one or more of the following findings, or associated relevant tumors: a. abnormal cerebrospinal fluid (CSF) b. neuroimaging or electrophysiological abnormalities. C. confirmatory test: positive neuronal autoantibodies. D. exclusion of other causes: a reasonable exclusion of other potential etiologies.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CASE | 2 months of enrollment
  The unabbreviated scale title is the clinical assessment scale for autoimmune encephalitis. The CASE includes a total score of 0-27.The higher the score, the worse the prognosis.

SECONDARY OUTCOMES:
CASE | 1 month of enrollment
  The unabbreviated scale title is the clinical assessment scale for autoimmune encephalitis. The CASE includes a total score of 0-27.The higher the score, the worse the prognosis.
mRS | 1 months, 2 months of enrollment
  The unabbreviated scale title is modified Rankin Scale. The mRS includes 0-6, and the higher the score, the worse the prognosis.
GCS | 1 months, 2 months of enrollment
  The unabbreviated scale title is Glasgow coma score. The GCS tested 3 components: eye opening response, verbal response and motor response, with a total score of 15. The lower the score, the more severe the brain damage and the deeper the degree of DOC.
Prognostic scores (CASE) | 6 months, 12 months of enrollment
  The unabbreviated scale title is the clinical assessment scale for autoimmune encephalitis. The CASE includes a total score of 0-27.The higher the score, the worse the prognosis.
Prognostic scores (mRS) | 6 months, 12 months of enrollment
  The unabbreviated scale title is modified Rankin Scale. The mRS includes 0-6, and the higher the score, the worse the prognosis.

IPD SHARING:
Plan to Share IPD: Undecided